CLINICAL TRIAL: NCT01681979
Title: WEUSRTP4850: Phase II: Asthma Treatment in Pregnancy and the Frequency of Adverse Pregnancy Outcomes
Brief Title: WEUSRTP4850: Phase II: ICS/LABA Use in Pregnancy and Outcomes
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114593; WEUSRTP4850 (Other: GSK); EPI40638 (Other: GSK)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Asthma
Keywords: fluticasone propionate; asthma; pregnancy; major congenital malformations
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with asthma during pregnancy: Women with asthma during pregnancy will be identified based on one of the following: 1) an asthma related medical code recorded anytime before the pregnancy start date and at least one prescription for an asthma medicine in the 6 months before the pregnancy start date or during pregnancy; 2) no asthma related medical code but at least 6 prescriptions for an asthma medicine in their record before the pregnancy start date, including one in the 6 months before the pregnancy start date or during pregnancy.
  Interventions: Drug: Fluticasone propionate (with and without concurrent salmeterol)

INTERVENTIONS:
Drug: Fluticasone propionate (with and without concurrent salmeterol) — Fluticasone propionate is an inhaled corticosteroid used for the treatment of asthma, often in combination with the long-acting β-agonist salmeterol. For the primary endpoint, exposure status will be determined based on the individual receiving a prescription for the drug of interest (fluticasone propionate or another inhaled corticosteroid) in the 2 weeks immediately before the LMP date or during the first trimester of pregnancy.
  Sensitivity analysis will be carried out categorising exposure based on mapping the duration of prescriptions based on the number of inhalers, number of puffs within an inhaler and the prescribed daily dose.

SUMMARY:
Asthma is reported to affect between 3-14% of pregnancies making asthma medicines one of the most commonly used classes of medicines during pregnancy. Maternal asthma and in particular poorly controlled asthma has been found to be associated with a number of adverse perinatal outcomes including preterm delivery, low birth weight and pre-eclampsia. At present little is known about the safety in humans of many anti-asthma medicines when used during pregnancy. As a result all inhaled corticosteroids, with the exception of budesonide which is category B, have an FDA pregnancy category C, indicative of the fact there are no adequate and well controlled studies in humans.

Fluticasone propionate is an inhaled corticosteroid used for the treatment of asthma, often in combination with the long-acting β-agonist salmeterol. Owing to small numbers of pregnancy exposures in the past, little is known about the safety of fluticasone propionate when used during pregnancy. A recent feasibility study, however, has shown that there are sufficient numbers of first trimester exposed pregnancies on the General Practice Research Database (GPRD) to allow the overall risk of major congenital malformations (MCMs) to be evaluated. This study also demonstrated that using data from the GPRD it is possible to determine an individual's exposure to anti-asthma medicines during pregnancy and to classify her treatment in terms of the British Thoracic Society treatment steps based on linked prescription and primary care data.

The aims of this study are to 1) evaluate the safety profile of fluticasone propionate (FP) compared with exposure to all other inhaled corticosteroids with all major congenital malformations combined as the primary endpoint, whilst taking into account potential confounders and exposure to other anti-asthma medicine; and 2) test the null hypothesis that exposure to fluticasone propionate during the first trimester of pregnancy is not associated with increased overall risk of all major congenital malformations when compared to the risk in those exposed to other inhaled corticosteroids during the first trimester of pregnancy.

The study will be a retrospective cohort study and will use data from the United Kingdom's General Practice Research Database (GPRD). The GPRD contains longitudinal medical records collected within UK primary care. All medical symptoms and diagnoses are recorded in the database, including those relating to pregnancy, in the form of Read Codes. In addition to coded data GPs have the option of recording un-coded comments ('free text'), such as more detailed descriptions of diagnoses or treatments along with information provided to them via hospital letters, referrals and discharge summaries.

As the recording of stillbirths, neonatal deaths and pre-term births on the GPRD has not been verified, a verification exercise will be carried out. This will involve requesting and reviewing free text comments for 100 stillbirths, 100 neonatal deaths and 100 pre-term births. Free text comments will be requested if they are associated with a medical code related to pregnancy, delivery, post natal visits, death, post mortem, hospital letters and other forms of communication. If the free text is not found to be informative we will send questionnaires to the woman's GP.

All outcomes will be identified and verified blinded to asthma treatment and severity levels.

ELIGIBILITY:
Inclusion Criteria:

* female patients whose pregnancy was registered on the GPRD and started and ended between 1 January 2000 and 31 December 2010
* Patients are considered to have asthma based on diagnosis and prescription codes

Exclusion Criteria:

* patients not registered with a practice contributing up-to-standard data to the GPRD for the 6 months before the start of pregnancy, throughout pregnancy and for the 3 months following the pregnancy end date.
* patients not 11-50 years of age on the pregnancy start date
* patients who experienced multiple birth (twins, triplets)
* patients with a medical code for a diagnosis of chronic obstructive pulmonary disease (COPD) or any other chronic respiratory condition (e.g. cystic fibrosis) recorded at anytime before the pregnancy end date

Ages: 11 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of all eligible pregnancies identified from the source population where the female is considered to have asthma. The source population will be all pregnancies identified on the GPRD that started and ended between 1 January 2000 and 31 December 2010.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
All major congenital malformations (MCMs) combined | 11 years (January 1, 2000 to December 31, 2010)

SECONDARY OUTCOMES:
Secondary outcomes associated with measures of asthma control, not drug exposures of interest including Spontaneous pregnancy losses, pre-term births, and Stillbirths and neonatal deaths. | 11 years (January 1, 2000 to December 31, 2010)
  Spontaneous pregnancy losses will be defined as losses that occurred > 24 wks gestation from the date of the first day of the last menstrual period (LMP) (identified based on the pregnancy algorithm). For pregnancy losses where the type of loss is unknown any free text comments associated with the code will be requested & reviewed. Pre-term births will be defined as a live birth delivered at <37 complete wks gestation from the date of the first day of the LMP (identified based on medical codes for a pre-term delivery in addition to gestational age & first day of LMP). Stillbirths =>24 wks.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline